CLINICAL TRIAL: NCT02943317
Title: A Phase 1/1b Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Clinical Activity of Defactinib in Combination With Avelumab in Epithelial Ovarian Cancer
Brief Title: Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Clinical Activity of Defactinib in Combination With Avelumab in Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated upon completion of escalation phase, prior to opening expansion cohorts
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-107
Record Dates: First submitted 2016-10-17; First posted 2016-10-24 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2018-07

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: VS-6063 (Experimental): Part A - Oral VS-6063 (defactinib) twice-daily (BID) continuously starting on Day 1 of Cycle 1.
  Interventions: Drug: Part A - VS-6063
- Part A: Avelumab (Experimental): Part A - avelumab IV treatment in 28-day cycles (10 mg/kg over approximately 1 hour on Days 1 and 15).
  Interventions: Drug: Part A - Avelumab

INTERVENTIONS:
Drug: Part A - VS-6063 — Part A - Oral VS-6063 (defactinib) twice-daily (BID) continuously starting on Day 1 of Cycle 1.
  Other Names: Defactinib
  Arms: Part A: VS-6063
Drug: Part A - Avelumab — Part A - avelumab IV treatment in 28-day cycles (10 mg/kg over approximately 1 hour on Days 1 and 15).
  Arms: Part A: Avelumab

SUMMARY:
This is a Phase 1/1b, open-label, multicenter, dose-escalation and dose expansion trial to evaluate the safety, efficacy, PK and PD of defactinib (VS-6063) in combination with avelumab in epithelial ovarian cancer.

DETAILED DESCRIPTION:
The study is comprised of 2 sequential parts: Part A (Dose Escalation of VS-6063) and Part B (Expansion).

In Part A (Dose Escalation), approximately 18 subjects will receive avelumab IV treatment in 28-day cycles (10 mg/kg over approximately 1 hour on Days 1 and 15) and oral defactinib twice-daily (BID) continuously starting on Day 1 of Cycle 1. Subject enrollment will proceed according to a standard 3+3 design. In the absence of dose-limiting toxicity (DLT), each subject will receive the study drug regimen for a minimum of 28 days (Cycle 1) and may continue to receive additional cycles of study treatment until disease progression has been documented or unacceptable toxicity or other treatment discontinuation criteria have been met. All subjects in a cohort must have completed at least 1 cycle of dosing before dose escalation involving new subjects entered into the next dose cohort can occur. Based on the safety and PK data obtained in the dose escalation portion of the study, the RP2D of the combination will be determined.

In Part B (Expansion), approximately 80 subjects will be enrolled and will receive avelumab IV treatment in 28-day cycles (10 mg/kg over approximately 1 hour on Days 1 and 15) and oral defactinib at the RP2D dose continuously starting on Day 1 of Cycle 1.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent before initiation of any study procedures.
2. Willing and able to participate in the trial and comply with all trial requirements.
3. Female subject aged ≥ 18 years.
4. Histologically or cytologically-confirmed recurrent or resistant (progression within 6 months following the last administered platinum based therapy or progression after subsequent therapy in previously relapsed subjects), stage III-IV epithelial ovarian, fallopian tube or peritoneal cancer subjects (according to American Joint Committee on Cancer/Union for International Cancer Control TNM and International Federation of Gynecology and Obstetrics Staging System, 7th edition) whose disease has progressed following adjuvant therapy or therapy for metastatic disease.
5. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
6. Confirmed availability of archived FFPE tumor tissue block, or a minimum of 15 slides. If archived FFPE tissue is not available, then fresh tumor sample may be obtained in accordance with local institutional practice for tumor biopsies.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1, measured within 72 hours before the start of treatment.
8. Predicted life expectancy of ≥ 3 months.
9. Adequate renal function with normal serum creatinine, or if creatinine above or below institutional normal range, a calculated glomerular filtration rate of ≥ 50 mL/min/1.73m2 (e.g., as calculated by the Cockcroft Gault formula) using actual body weight; if subject has body mass index > 30 kg/m2, lean body weight must be used.
10. Adequate hepatic function (total bilirubin ≤ 1.5 × upper limit of normal [ULN] for the institution; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN.
11. Adequate bone marrow function (hemoglobin [Hb] ≥ 9.0 g/dL [subjects may be transfused to Hb ≥ 9.0 g/dL]; platelets ≥ 100 × 109cells/L; absolute neutrophil count [ANC] ≥ 1.5 × 109 cells/L without the use of hematopoietic growth factors).
12. Corrected QT interval (QTc) < 470 msec (as calculated by the Fridericia correction formula [QTcF]).
13. Negative pregnancy test within 72 hours prior to the first dose of protocol therapy for women of childbearing potential. Must be willing to use effective contraception for 30 days before the first study drug administration, for the duration of trial participation and at least for 60 days after stopping trial participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician must be informed immediately.

Exclusion Criteria:

1. Concurrent anticancer treatment, major surgery or use of any investigational drug within 28 days or 5 half-lives, whichever is shorter, before the start of trial treatment; palliative radiation therapy is allowed if > 21 days before planned first dose of study drugs and any toxicity is ≤ Grade 1.
2. Concurrent systemic therapy with immunosuppressive agents; use of hormonal agents within 7 days before the start of trial treatment. Note: subjects receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before the first dose of avelumab. Subjects receiving immunosuppressive agents (such as corticosteroids) for any reason should be tapered off these drugs before initiation of the study treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to ≤ 10 mg prednisone daily). Steroids with no or minimal systemic effect (topical, inhalation) are allowed.
3. Prior treatment with a drug of the focal adhesion kinase (FAK) inhibitor class.
4. Prior therapy with specific antibody/drug targeting immune or coregulatory or costimulatory proteins (such as checkpoints e.g., PD-1 or PD L1, 4-1BB, OX40 or CTLA-4 antibodies).
5. Receipt of any organ transplantation including autologous or allogeneic stem-cell transplantation.
6. Uncontrolled brain metastases (Stable brain metastases either treated or being treated with a stable dose of anticonvulsants, with no dose change within 28 days before enrollment, will be allowed.).
7. Women who are pregnant or breastfeeding.
8. Any evidence of serious active infections; any infections being treated must complete antibiotic therapy at least 7 days before planned first dose.
9. Active or history of any autoimmune disease (subjects with diabetes type 1, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible).
10. Current acute or chronic colitis, inflammatory bowel disease, pneumonitis or pulmonary fibrosis.
11. Known severe hypersensitivity reactions to monoclonal antibodies; any history of anaphylaxis or uncontrolled asthma.
12. Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months before study treatment, New York Heart Association Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease or cardiac amyloidosis.
13. Known history of stroke or cerebrovascular accident within 6 months before enrollment.
14. Known infection with human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS) (testing not required).
15. Active hepatitis B or C (testing required).
16. Known history of Gilbert's Syndrome.
17. Other uncontrolled or poorly controlled intercurrent illness (e.g., involving the renal, hepatic, neurologic, dermatologic, pulmonary, endocrine systems) or psychiatric illness/social situations that would limit compliance with study requirements, place the subject at undue risk or confound interpretation of safety or other data.
18. Gastrointestinal (GI) condition that could interfere with the swallowing or absorption of defactinib.
19. History of upper GI bleeding, ulceration or perforation within 6 months before the first dose of defactinib.
20. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
21. Previous malignant disease other than the target malignancy to be investigated in this trial within the last 3 years, with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ. Any prior cancer must not be getting active treatment and must be in continuous complete remission for at least 3 years.
22. Persisting toxicity related to prior therapy > Grade 1 National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 (NCI-CTCAE v4.03); however, sensory neuropathy ≤ Grade 2 is acceptable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants taking defactinib in combination with avelumab with Adverse Events as a Measure of Safety and Tolerability | Up to 90 days after last dose
maximum tolerated dose (MTD) of defactinib in combination with avelumab (Part A) | From start of treatment to end of Cycle 1 (28 days)
best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Part B) | From start of treatment, assessed up to 52 weeks

SECONDARY OUTCOMES:
time to treatment response disease control | 12, 24, 36, and 52 weeks
best overall response according to immune-related response evaluation criteria in solid tumors (irRECIST) | From start of treatment, assessed up to 52 weeks
immune related progression-free survival (irPFS) time according to irRECIST and RECIST v1.1 | From start of treatment until first documented progression or death, whichever comes first, assessed up to 52 weeks
progression-free survival (PFS) time according to irRECIST and RECIST v1.1 | From start of treatment until first documented progression or death, whichever comes first, assessed up to 52 weeks
overall Survival (OS) | From start of treatment until death, assessed up to 52 weeks
duration of response (DOR) according to irRECIST and RECIST v1.1 | From start of treatment until first documented progression, assessed up to 52 weeks
plasma concentration of avelumab and defactinib | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (5):
- United States (5):
  - Florida Cancer Specialists & Research Institute (FCS), Sarasota, Florida
  - Dana Farber Cancer Instiyute, Boston, Massachusetts
  - Stephenson Cancer Center (University of Oklahoma), Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided